CLINICAL TRIAL: NCT05678504
Title: The Effect of Using Blood Vessel Imaging Device on Pain and Satisfaction Level During the Phlebotomy Procedure
Brief Title: The Process of Blood Collection With a Vascular Imaging Device
Acronym: VID
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, özlem doğu, Assoc. Dr., Sakarya University
Other Study IDs: Blood vessel imaging device
Record Dates: First submitted 2022-10-10; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Phlebotomy
Keywords: Phlebotomy; blood vessel imaging device; pain; satisfaction
MeSH Terms: conditions — Pain; Personal Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Application Group: * Filling out the pre-initiative volunteering form and sociodemographic data
  * Preparation of the individual for the transaction
  * Monitoring the vein with a vein imaging device and operating a stopwatch
  * Implementation of the initiative
  * Stopping the stopwatch at the end of the process
  * Application of VAS Pain and VAS satisfaction Scale
  Interventions: Device: The phlebotomy procedure
- Control Group: * Filling out the pre-initiative volunteering form and sociodemographic data
  * Preparation of the individual for the transaction
  * Starting routine blood collection and starting the stopwatch
  * Implementation of the initiative
  * Stopping the stopwatch at the end of the process
  * Application of VAS Pain and VAS satisfaction Scale

INTERVENTIONS:
Device: The phlebotomy procedure — The process of blood collection with a vascular imaging device
  Groups: Application Group

SUMMARY:
The study was planned to determine the effect of using a blood vessel imaging device (VID) and venous blood collection procedure on the pain and satisfaction level of the individual during phlebotomy. The randomized controlled experimental design study was carried out in a blood collection unit in a training and research hospital between 1-15 April 2022. The study sample was calculated as 100 people by power analysis and the method of drawing lots was applied to the groups. Data were collected using the patient identification form, visual analogue scale (VAS), and pain and satisfaction scales.

DETAILED DESCRIPTION:
The population of the study consisted of adult individuals who benefited from polyclinic services and applied to the blood collection unit between the specified dates in a single center.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-65,
* Who wanted peripheral vascular access,
* Volunteered to participate in the study,
* Did not have any pain complaints,
* Did not take analgesics in the last 12 hours,
* Could be contacted,
* Did not have obesity, dehydration, peripheral oedema, or a cancer diagnosis and did not need emergency intervention.

Exclusion Criteria:

* Those who do not meet the criteria for admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 application grup 50 control grup
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
The effect of using a blood vessel imaging device on the pain of the phlebotomy procedure | one month
  Blood vessel imaging device effective pain level

SECONDARY OUTCOMES:
The effect of using a blood vessel imaging device on satisfaction level during the phlebotomy procedure | one month
  Blood vessel imaging device effective satisfaction level

CONTACTS AND LOCATIONS:
Overall Officials: özlem doğu, assoc. dr, Principal Investigator — Sakarya University
Locations (1):
- Sakarya training and research hospital, Sakarya, Adapazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guillon P, Makhloufi M, Baillie S, Roucoulet C, Dolimier E, Masquelier AM. Prospective evaluation of venous access difficulty and a near-infrared vein visualizer at four French haemophilia treatment centres. Haemophilia. 2015 Jan;21(1):21-6. doi: 10.1111/hae.12513. Epub 2014 Oct 21. PMID 25335191
- [Background] Amick AE, Feinsmith SE, Sell J, Davis EM, Wayne DB, Feinglass J, Barsuk JH. Ultrasound-Guided Peripheral Intravenous Catheter Insertion Training Reduces Use of Midline Catheters in Hospitalized Patients With Difficult Intravenous Access. J Patient Saf. 2022 Apr 1;18(3):e697-e703. doi: 10.1097/PTS.0000000000000910. PMID 34570003
- [Background] Revill SI, Robinson JO, Rosen M, Hogg MI. The reliability of a linear analogue for evaluating pain. Anaesthesia. 1976 Nov;31(9):1191-8. doi: 10.1111/j.1365-2044.1976.tb11971.x. PMID 1015603
- [Result] Kim K, Jeong HW, Lee Y. Performance Evaluation of Dorsal Vein Network of Hand Imaging Using Relative Total Variation-Based Regularization for Smoothing Technique in a Miniaturized Vein Imaging System: A Pilot Study. Int J Environ Res Public Health. 2021 Feb 6;18(4):1548. doi: 10.3390/ijerph18041548. PMID 33561967
- [Result] Zhang Z, Wang X, Zhang L, Lou X, Su X, Wang X, Sun F, He X. Infrared Vein Imaging for Insertion of Peripheral Intravenous Catheter for Patients Requiring Isolation for Severe Acute Respiratory Syndrome Coronavirus 2 Infection: A Nonrandomized Clinical Trial. J Emerg Nurs. 2022 Mar;48(2):159-166. doi: 10.1016/j.jen.2021.10.001. Epub 2021 Oct 12. PMID 35115182
- [Result] Aulagnier J, Hoc C, Mathieu E, Dreyfus JF, Fischler M, Le Guen M. Efficacy of AccuVein to facilitate peripheral intravenous placement in adults presenting to an emergency department: a randomized clinical trial. Acad Emerg Med. 2014 Aug;21(8):858-63. doi: 10.1111/acem.12437. PMID 25176152
- [Result] Eren H, Caliskan N. Effect of a Vein Imaging Device and of Fist Clenching on Determination of an Appropriate Vein and on Catheter Placement Time in Patients Receiving Chemotherapy: A Randomized Controlled Trial. Cancer Nurs. 2022 Mar-Apr 01;45(2):105-112. doi: 10.1097/NCC.0000000000000931. PMID 33654007
- [Result] Morata L, Bowers M. Ultrasound-Guided Peripheral Intravenous Catheter Insertion: The Nurse's Manual. Crit Care Nurse. 2020 Oct 1;40(5):38-46. doi: 10.4037/ccn2020240. PMID 33000131
- [Result] Skulec R, Callerova J, Vojtisek P, Cerny V. Two different techniques of ultrasound-guided peripheral venous catheter placement versus the traditional approach in the pre-hospital emergency setting: a randomized study. Intern Emerg Med. 2020 Mar;15(2):303-310. doi: 10.1007/s11739-019-02226-w. Epub 2019 Nov 7. PMID 31701317
- [Result] Yilmaz Kurt F, Aytekin Ozdemir A, Atay S. The Effects of Two Methods on Venipuncture Pain in Children: Procedural Restraint and Cognitive-Behavioral Intervention Package. Pain Manag Nurs. 2020 Dec;21(6):594-600. doi: 10.1016/j.pmn.2019.09.002. Epub 2019 Oct 15. PMID 31628067
- See also: Zhu, Q., Zhang, Z., Liu, N., & Sun, H. (2015). Near infrared hand vein image acquisition and extraction algorithm. Optics, 126(24), 5682-5687. — https://www.infona.pl/resource/bwmeta1.element.elsevier-1d4b899a-3c22-30c7-a988-a5990180d27b
- See also: CURRENT APPROACH TO PEDIATRIC VASCULAR ACCESS APPLICATIONS: VESSEL VISUALIZATION TECHNIQUE — http://journal.acibadem.edu.tr/tr/download/article-file/1701903